CLINICAL TRIAL: NCT00516503
Title: The Use of Topical Baclofen, Amitriptyline HCI, and Ketamine (BAK) in a PLO Gel vs. Placebo for the Treatment of Chemotherapy Induced Peripheral Neuropathy: A Phase III Randomized Double-Blind Placebo Controlled Study
Brief Title: Baclofen-Amitriptyline Hydrochloride-Ketamine Gel in Treating Peripheral Neuropathy Caused by Chemotherapy in Patients With Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCCTG-N06CA; NCI-2011-01768 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000560732 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2007-08-14; First posted 2007-08-15 (Estimated); Results first posted 2017-08-24 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-07

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Lymphoproliferative Disorder; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms; Neurotoxicity; Pain; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Lymphoproliferative Disorders; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Neurotoxicity Syndromes; Pain | interventions — Baclofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients apply 1 spoonful of baclofen-amitriptyline hydrochloride-ketamine gel> topically to each> area of pain,> numbness,> and/or tingling> on the> feet and/or hands twice daily> for> 4 weeks.
  Interventions: Drug: baclofen/amitriptyline/ketamine gel
- Arm II (Placebo Comparator): Patients apply 1 spoonful of placebo gel topically to each area of pain, numbness, and/or tingling on the feet and/or hands twice daily for 4 weeks.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: baclofen/amitriptyline/ketamine gel — Applied topically
  Arms: Arm I
Other: placebo — Applied topically
  Arms: Arm II

SUMMARY:
RATIONALE: Baclofen-amitriptyline-ketamine (BAK) gel may lessen peripheral neuropathy caused by chemotherapy. It is not yet known whether BAK gel is more effective than a placebo in treating peripheral neuropathy caused by chemotherapy .

PURPOSE: This randomized phase III trial is studying BAK gel to see how well it works compared with a placebo in treating peripheral neuropathy caused by chemotherapy in patients with cancer.

DETAILED DESCRIPTION:
OBJECTIVES Primary

* Compare the effectiveness of baclofen-amitriptyline hydrochloride-ketamine (BAK) gel versus placebo, in terms of improving sensory neuropathy, in cancer patients with chemotherapy-induced peripheral neuropathy> Secondary>
* Compare motor and autonomic symptoms and functioning, mood states, pain, and peripheral neuropathy in these patients.
* Assess the adverse event profile of topical BAK gel.
* Explore whether topical BAK gel is absorbed systemically. OUTLINE: Patients are stratified according to neurotoxic chemotherapy (active vs non-active), current use of opioids or oral pain medications (yes vs no), pain rating (4-7 vs 8-10), and prior ineffective pharmacologic treatment for peripheral neuropathy (yes vs no). Patients are randomized to 1 of 2 treatment arms.
* Arm I: Patients apply 1 spoonful of baclofen-amitriptyline hydrochloride-ketamine gel topically to each area of pain, numbness, and/or tingling on the feet and/or hands twice daily for 4 weeks.
* Arm II: Patients apply 1 spoonful of placebo gel topically to each area of pain, numbness, and/or tingling on the feet and/or hands twice daily for 4 weeks.

Some patients in both arms may choose to continue on the active gel or, if on placebo, begin the active gel for an additional 8 weeks off study. Patients complete health, pain, mood, and quality of life questionnaires at baseline and periodically during study. Patients also record adverse symptoms weekly in a Symptom Experience Diary.

ELIGIBILITY:
DISEASE CHARACTERISTICS:>

* Diagnosis of cancer>
* Received or currently receiving neurotoxic chemotherapy including, but not limited to, taxanes (e.g., paclitaxel or docetaxel); platinum-based compounds (e.g., carboplatin, cisplatin, or oxaliplatin); vinca alkaloids (e.g., vincristine or vinblastine); or other neurotoxic chemotherapy agents (e.g., bortezomib, lenalidomide, or thalidomide)>
* Must have pain or symptoms of peripheral neuropathy attributable to chemotherapy for ≥ 1 month>

  * Neuropathy is limited to either hands and/or feet where gel can be applied>
  * Neuropathic pain score of ≥ 4 out of 10 on the numbness/tingling/pain numeric analogue scale>
* No pre-existing or history of peripheral neuropathy due to any cause other than chemotherapy (e.g., diabetes, alcohol, toxin, heredity)> PATIENT CHARACTERISTICS:>
* ECOG performance status 0-2>
* Life expectancy ≥ 4 months>
* Creatinine ≤ 1.5 times upper limit of normal>
* Not pregnant or nursing>
* No ability to bear children defined by 1 of the criteria:>

  * Menopausal (12 months and no menstrual period if natural menopause)>
  * Underwent a hysterectomy and/or oophorectomy>
  * Permanent surgical sterilization (tubal ligation)>
* Fertile patients must use effective contraception>
* Able to complete questionnaires independently or with assistance>
* Able to sign informed consent and understand the nature of a placebo-controlled trial>
* No history of an allergic reaction to baclofen, amitriptyline hydrochloride, and/or ketamine>
* No diagnosis of any New York Heart Association class I-IV congestive heart failure>
* No diagnosis of coronary artery disease including, but not limited to, myocardial infarction, within the past 5 years>
* No other medical condition that, in the opinion of the treating physician or allied health professional, would make this clinical trial unreasonably hazardous for the patient>
* No skin abnormalities at the intended application sites (hands and feet) of study gel (i.e., skin breakdown)> PRIOR CONCURRENT THERAPY:>
* See Disease Characteristics>
* More than 30 days since prior anticonvulsants, tricyclic antidepressants, monoamine oxidase inhibitor, or other neuropathic pain medication (e.g., carbamazepine, phenytoin, valproic acid, gabapentin, lamotrigine, topical lidocaine patch or gel, capsaicin cream, or amifostine)>

  - Patients treated with any of these agents for peripheral neuropathy for ≤ 1 week during the past 30 days are eligible provided they are no longer taking the agent>
* More than 5 years since prior percutaneous transluminal coronary angioplasty or coronary artery bypass graft>

  - Prior heart valve replacement surgery allowed provided patient has fully recovered from the surgery>
* No concurrent use of study agents other than as specified in the trial>

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2008-02; Primary Completion 2009-04 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra Barton, RN, PhD, AOCN, FAAN, Study Chair — Mayo Clinic
Locations (165):
- United States (165):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Moline, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Bettendorf, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Immanuel St. Joseph's, Mankato, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - North Coast Cancer Care - Clyde, Clyde, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center and Children's Hospital, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Guthrie Cancer Center at Guthrie Clinic Sayre, Sayre, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Mercy Hospital at Wilkes-Barre, Wilkes-Barre, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Franciscan Skemp Healthcare - La Crosse Campus, La Crosse, Wisconsin

REFERENCES:
- [Result] Wolf SL, Barton DL, Qin R, Wos EJ, Sloan JA, Liu H, Aaronson NK, Satele DV, Mattar BI, Green NB, Loprinzi CL. The relationship between numbness, tingling, and shooting/burning pain in patients with chemotherapy-induced peripheral neuropathy (CIPN) as measured by the EORTC QLQ-CIPN20 instrument, N06CA. Support Care Cancer. 2012 Mar;20(3):625-32. doi: 10.1007/s00520-011-1141-9. Epub 2011 Apr 12. PMID 21479990
- [Result] Barton DL, Wos EJ, Qin R, Mattar BI, Green NB, Lanier KS, Bearden JD 3rd, Kugler JW, Hoff KL, Reddy PS, Rowland KM Jr, Riepl M, Christensen B, Loprinzi CL. A double-blind, placebo-controlled trial of a topical treatment for chemotherapy-induced peripheral neuropathy: NCCTG trial N06CA. Support Care Cancer. 2011 Jun;19(6):833-41. doi: 10.1007/s00520-010-0911-0. Epub 2010 May 25. PMID 20496177
- [Result] Barton DL, Wos E, Qin R, et al.: A randomized controlled trial evaluating a topical treatment for chemotherapy-induced neuropathy: NCCTG trial N06CA. [Abstract] J Clin Oncol 27 (Suppl 15): A-9531, 2009.
- [Result] Wolf SL, Qin R, Barton DL, et al.: Relationship of sensory symptoms and motor function in patients with chemotherapy-induced peripheral neuropathy (CIPN) utilizing the EORTC QLQ CIPN20: NCCTG study N06CA. [Abstract] J Clin Oncol 27 (Suppl 15): A-9587, 2009.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two-hundred eight patients were enrolled to this study. Five patients cancelled prior to initiating protocol treatment and were therefore this study was analyzed using 203 remaining patients.
Groups:
- Baclofen-amitriptyline Hydrochloride-ketamine: Patients apply 1 spoonful of baclofen-amitriptyline hydrochloride-ketamine gel topically to each area of pain, numbness, and/or tingling on the feet and/or hands twice daily for 4 weeks. Baclofen/amitriptyline/ketamine gel: Applied topically.
- Placebo: Patients apply 1 spoonful of placebo gel topically to each area of pain, numbness, and/or tingling on the feet and/or hands twice daily for 4 weeks. Placebo: Applied topically
Period: Overall Study
Arm/Group | Baclofen-amitriptyline Hydrochloride-ketamine | Placebo
Started | 101 | 102
Completed | 101 | 102
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Baclofen-amitriptyline Hydrochloride-ketamine | Placebo | Total
Number analyzed (Participants) | 101 | 102 | 203
Age, Continuous [Median (Full Range); unit: years] | 59.5 [41 to 83] | 62 [31 to 86] | 61 [31 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 60 | 126
  Male | 35 | 42 | 77
Region of Enrollment [Number; unit: participants]
  United States | 101 | 102 | 203

OUTCOME MEASURES:

1. Primary Outcome: Total Sensory Neuropathy as Measured by the European Organization for Research and Treatment of Cancer [EORTC] Quality of Life [QLQ] - Chemo-induced Peripheral Neuropathy [CIPN20]
Description: The scoring algorithm for the parent instrument, the EORTC QLQ-C30, was applied for linearly converting items and subscales of CIPN-20 to 0-100 scales so that a high score corresponds to better condition or less symptom. The primary analysis was the change in sensory neuropathy subscale of the CIPN-20 from baseline to week 4. The area under the curve (AUC) from baseline to week 4 was calculated for each patient's sensory neuropathy score. The average AUC for the placebo arm was compared to the average AUC for the topical amitriptyline HCl/ baclofen/ ketamine arm using a Wilcoxon rank sum test.
Time Frame: From baseline to 4 weeks
Population: There were 26 participants in the BAK arm and 27 in the placebo arm who did not provide primary endpoint data. In the BAK arm, 11 refused due to experiencing an adverse event and 15 refused for non-specified reasons. In the placebo arm, eight refused due to an adverse event, one patient died, and 18 refused for non-specified reasons.
Measure: Mean (Standard Deviation); unit: (units on a scale) * week
Arm/Group | Baclofen-amitriptyline Hydrochloride-ketamine | Placebo
Number analyzed (Participants) | 75 | 75
(units on a scale) * week | 61.0 (16.22) | 60.9 (17.9)
Statistical Analysis 1: Comparison: Baclofen-amitriptyline Hydrochloride-ketamine vs Placebo; Test type: Superiority or Other; p = 0.90, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Motor Neuropathy as Measured by the EORTC QLQ-CIPN20 at Baseline and Week 4
Description: The scoring algorithm for the parent instrument, the EORTC QLQ-C30, was applied for linearly converting items and subscales of CIPN-20 to 0-100 scales so that a high score corresponds to better condition or less symptom. The secondary analysis was to compare changes from baseline at 4 weeks for the motor neuropathy subscale of the CIPN-20. To analyze this endpoint, the area under the curve (AUC) from baseline to week 4 was calculated for each patient's motor neuropathy score. The average AUC for the placebo arm was compared to the average AUC for the topical amitriptyline HCl/ baclofen/ ketamine arm using a Wilcoxon rank sum test.
Time Frame: From Baseline to week 4
Population: There were 26 participants in the BAK arm and 27 in the placebo arm who did not provide primary endpoint data. In the BAK arm, 11 refused due to experiencing an adverse> event and 15 refused for non-specified reasons. In the placebo arm, eight refused due to an> adverse event, one patient died, and 18 refused for non-specified reasons.
Measure: Mean (Standard Deviation); unit: (units on a scale)* week
Arm/Group | Baclofen-amitriptyline Hydrochloride-ketamine | Placebo
Number analyzed (Participants) | 75 | 75
(units on a scale)* week | 69.2 (17.15) | 70.1 (19.48)
Statistical Analysis 1: Comparison: Baclofen-amitriptyline Hydrochloride-ketamine vs Placebo; Test type: Superiority or Other; p = 0.50, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Autonomic Symptoms and Functioning as Measured by the EORTC QLQ-CIPN20 at Baseline and Week 4
Description: The scoring algorithm for the parent instrument, the EORTC QLQ-C30, was applied for linearly converting items and subscales of CIPN-20 to 0-100 scales so that a high score corresponds to better condition or less symptom. The secondary analysis was to compare changes from baseline at 4 weeks for the autonomic neuropathy subscale of the CIPN-20. To analyze this endpoint, the area under the curve (AUC) from baseline to week 4 was calculated for each patient's motor neuropathy score. The average AUC for the placebo arm was compared to the average AUC for the topical amitriptyline HCl/ baclofen/ ketamine arm using a Wilcoxon rank sum test.
Time Frame: Up to 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: (units on a scale)*week
Arm/Group | Baclofen-amitriptyline Hydrochloride-ketamine | Placebo
Number analyzed (Participants) | 75 | 75
(units on a scale)*week | 85.0 (15.47) | 86.8 (15.03)
Statistical Analysis 1: Comparison: Baclofen-amitriptyline Hydrochloride-ketamine vs Placebo; Test type: Superiority or Other; p = 0.50, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Mood States and Total Mood Disturbance as Measured by the Profile of Mood States (POMS)
Description: Each mood scale (0 - 100, higher is better mood) will be analyzed as an endpoint along with the total mood disturbance score.
Time Frame: At 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baclofen-amitriptyline Hydrochloride-ketamine | Placebo
Number analyzed (Participants) | 101 | 102
units on a scale
  POMS Tension-Anxiety Subscale | 83.2 (17.09) | 83.0 (15.73)
  POMS VA Subscale | 31.1 (18.42) | 33.0 (19.61)
  POMS Anger-Hostility Score | 87.8 (14.48) | 87.7 (12.98)
  POMS Confusion-Bewilderment | 76.9 (17.58) | 77.9 (11.75)
  POMS Depression-Dejection Score | 86.4 (16.09) | 85.8 (15.23)
  POMS Fatigue-Inertia Score | 67.2 (21.69) | 63.6 (22.22)
  Mean POMS Score | 71.5 (13.27) | 71.8 (13.14)

5. Secondary Outcome: Pain Severity and Interference as Measured by the Brief Pain Inventory (BPI) at Baseline and Week 4
Description: Pain severity, defined by the four items addressing worst, least, and average pain and pain right now as measured by the BPI will be analyzed identical to the primary endpoint. Additionally, total pain interference as measured by the BPI will be transformed onto a 0-100 ( higher is less pain) point scale. The area under the curve (AUC) from baseline to week 4 was calculated for each patient's score. The average AUC for the placebo arm and the topical amitriptyline HCl/ baclofen/ ketamine arm are reported.
Time Frame: Up to 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale * week
Arm/Group | Baclofen-amitriptyline Hydrochloride-ketamine | Placebo
Number analyzed (Participants) | 101 | 102
units on a scale * week
  Worst Pain | 58.1 (25.48) | 58.7 (27.39)
  Least Pain | 78.0 (20.28) | 77.3 (22.01)
  Average Pain | 66.4 (21.99) | 65.4 (24.55)
  BPI Total Interference | 76.5 (20.16) | 77.3 (21.16)

6. Secondary Outcome: Numbness, Tingling, and Pain as Measured by the Peripheral Neuropathy Questionnaire at Baseline and Weekly for 4 Weeks
Description: The Peripheral Neuropathy Questionnaire was used to analyze this endpoint. Patient neuropathy symptoms were scored on a 0 - 100 scale (higher score represents less symptomatic). The area under the curve (AUC) from baseline to week 4 was calculated for each patient's score. The average AUC for the placebo arm and the topical amitriptyline HCl/ baclofen/ ketamine arm are reported.
Time Frame: Up to 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale * week
Arm/Group | Baclofen-amitriptyline Hydrochloride-ketamine | Placebo
Number analyzed (Participants) | 101 | 102
units on a scale * week | 172.6 (82.09) | 175.7 (85.38)

7. Secondary Outcome: Adverse Event Profile of Topical Amitriptyline HCl/ Baclofen/Ketamine > Frequency and Severity of Adverse Events Reported by the Patient in the > Symptom Experience Diary and Evaluated Through Clinical Assessment by NCI CTCAE v3.0
Description: Frequency and severity of adverse events reported by patients in weekly diary and evaluated through clinical assessment by NCI CTCAE v3.0. The number of patients reporting grade 3 or higher events are reported in this outcome measure. For a full list of all events, please refer to the Adverse Events section of this report.
Time Frame: Up to 4 weeks
Population: All patients that were assessed for adverse events are used in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Baclofen-amitriptyline Hydrochloride-ketamine | Placebo
Number analyzed (Participants) | 101 | 102
Participants
  Grade 3+ Adverse Event | 8 | 5
  Grade 4+ Adverse Event | 1 | 1

ADVERSE EVENTS:
Arm/Group | Baclofen-amitriptyline Hydrochloride-ketamine | Placebo
Serious Adverse Events (participants affected / at risk) | 1/101 | 1/102
Other Adverse Events (participants affected / at risk) | 48/101 | 45/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baclofen-amitriptyline Hydrochloride-ketamine (N=101) | Placebo (N=102)
Disease progression (General disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baclofen-amitriptyline Hydrochloride-ketamine (N=101) | Placebo (N=102)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (5)
Constipation (Gastrointestinal disorders) | 24 (62) | 28 (71)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 18 (55) | 23 (55)
Ileal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (4)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Bladder infection (Infections and infestations) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (2) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 2 (2)
Syncope vasovagal (Nervous system disorders) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 5 (5) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 16 (26) | 12 (25)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No